CLINICAL TRIAL: NCT04803487
Title: Robotic Cholecystectomy Using the Newly Developed Chinese Robotic Surgical System-Micro Hand S: A Controlled, Randomized, Prospective Clinical Study
Brief Title: Robotic Cholecystectomy Using the Chinese Micro Hand S Robot: A Controlled, Randomized, Prospective Clinical Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Haitao Niu, MD, Professor Haitao Niu (The department of Urology), The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SDWG-NST600S-CT
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Cholecystitis; Gallstone
Keywords: Surgical robot; Robot-assisted cholecystectomy
MeSH Terms: conditions — Cholecystitis; Gallstones

STUDY DESIGN:
Intervention Model Description: random controlled trial
Who Masked: Participant
Masking Description: single-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Micro Hand S robot group (Experimental): 41 patients were randomly allocated in the Micro Hand S robot group and cholecystectomy was performed using the Micro Hand S robot.
  Interventions: Other: robot-assisted cholecystectomy
- the da Vinci robot group (Other): 41 patients were randomly allocated in the da Vinci robot group and cholecystectomy was performed using the da Vinci robot.
  Interventions: Other: robot-assisted cholecystectomy

INTERVENTIONS:
Other: robot-assisted cholecystectomy — cholecystectomy was performed for patients using the Chinese Micro Hand S surgical robot.
  Arms: the Micro Hand S robot group
Other: robot-assisted cholecystectomy — cholecystectomy was performed for patients using the da Vinci surgical robot.
  Arms: the da Vinci robot group

SUMMARY:
A single-blinded, prospective randomized parallel controlled clinical trial was designed and conducted from December 2019 to November 2020. 82 patients with a gallstone, gallbladder polyp and other benign gallbladder diseases were enrolled in this study. Finally, 82 patients were randomly divided into the Micro Hand S surgical robot group and the da Vinci surgical robot group. Standard robot-assisted transabdominal cholecystectomy was conducted using the Micro Hand S robot or the da Vinci robot. The success rate of operation, assembly time, operation time, intraoperative hemorrhage, time to first flatus, postoperative pain, comprehensive complication index, resident time and patient satisfaciton were recorded. The aim of the study is to determine whether the newly developed Chinese Micro Hand S surgical robot results in non-inferiority outcomes in cholecystectomy compared with the prevalent da Vinci robot.

DETAILED DESCRIPTION:
Objective: To determine whether the newly developed Chinese Micro Hand S surgical robot results in non-inferiority outcomes in cholecystectomy compared with the prevalent da Vinci robot.

Design: A single-blinded, prospective randomized parallel controlled clinical trial was designed and conducted from December 2019 to November 2020. The study was conducted in an academic hospital. 82 patients with a gallstone, gallbladder polyp and other benign gallbladder diseases were enrolled in this study. Finally, 82 patients were randomly divided into the Micro Hand S surgical robot group and the da Vinci surgical robot group.

Interventions: Standard robot-assisted transabdominal cholecystectomy was conducted using the Micro Hand S robot or the da Vinci robot.

Main outcomes and measures: The main outcome was the success rate of operation. Surgical success was defined as that the surgical procedures were completed by the experimental or control product without transferring to non-robotic surgery. Secondary outcomes included assembly time, operation time, intraoperative hemorrhage, time to first flatus, postoperative pain, comprehensive complication index, resident time and patient satisfaction.

Background:

Cholecystectomy is one of the most common operations in general surgery, with about half a million patients getting cholecystectomy each year in the United States. In the 1990s, minimally invasive surgery (MIS), as a new technology, greatly improved the traditional open abdominal surgery, of which defects are known as the big wound and long time to recover. Today, nearly 90% of cholecystectomy are performed laparoscopically. Previous studies have shown that laparoscopic cholecystectomy may reduce postoperative pain, shorten the hospital stay, and save the overall cost in hospital, which has become the standard operation for the treatment of gallbladder disease. In recent years, robot-assisted laparoscopic surgery has become more and more widely used in general surgery because of its advantages of 3D visions, high magnification, tremor suppression, and precise manipulation. According to a reported retrospective study, the da Vinci robot-assisted cholecystectomy showed excellent operation security, which can achieve the same therapeutic effect as the conventional laparoscopic cholecystectomy. But studies also reported that the increased cost may be the main problem of the da Vinci robot-assisted cholecystectomy.

The Micro Hand S surgical robot is a new generation of Chinese independently developed surgical robot system. Apart from the flexibility and intelligence in operation manipulation, the Micro Hand S surgical robot also has the advantages of small size, portable equipment, low maintenance costs and outstanding equipment compatibility. After initial preclinical trials, the Micro Hand S surgical robot has been successfully applied in clinic, and proved security and feasibility in various gastrointestinal surgery.

Since 2019, investigators in this group have designed and taken up research to assist laparoscopic cholecystectomy with the Micro Hand S surgical robot, which is noted as a prospective, randomized, single-blind, and parallel controlled clinical trial. The primary purpose of this study is to determine whether the newly developed Chinese Micro Hand S surgical robot results in non-inferiority outcomes in cholecystectomy compared with the prevalent da Vinci robot.

Method:

The study was designed as a single-blind prospective randomized clinical trial since it is inevitable for the surgeon to know what kind of robot to use during the operation. After obtaining the approval of the Ethics Review Committee and other relevant institutions of the Affiliated Hospital of Qingdao University, a total of 82 patients were included in this study from December 2019 to November 2020. Finally, 82 patients were randomly divided into the Micro Hand S robot group and the da Vinci robot group. All enrolled patients were fully informed and signed the informed consent. Patients were randomly assigned to each group in a 1:1 ratio, and information of the grouping and intervention measures were not available to patients. Patients of each group were matched for age, sex, body mass index (BMI), and complications to reduce confounding intervention factors.

Surgical procedure:

The patient was placed in the supine position after general anesthesia. The Veress needle was inserted at 2cm below the umbilicus (point A) to establish the CO2 artificial pneumoperitoneum. A 12mm trocar was inserted into the abdominal cavity and the pneumoperitoneum tube was connected to the trocar. The intra-abdominal pressure was set at 11-13mmHg, and then the preheated three-dimensional laparoscope and cold-light source were placed into the abdominal cavity through the trocar. Then a thorough examination was taken on the intended trocar points and the surgical area. After adjusting the patient with a Trendelenburg position inclined to the left, 10.5mm magnetic trocars were respectively placed at 2-3cm medial side of the right anterior axillary line, 8-10cm below the costal margin (point B); and 2-3cm below the costal margin of the left mid-clavicular line (point C); and were connected to the robotic arms No. 1 and 2. Besides, a 10mm trocar were placed at point D (lateral inferior of the line connecting point A and C) as the auxiliary channel. The surgeon held the neck of the gallbladder or Hartmann's Pouch with bipolar forceps, and pulled the neck to the right upper to open the serosal layer of the cystic duct. The cystic duct and the cystic artery were then separated by blunt dissection so as to distinguish the common bile duct, hepatic common bile duct, and cystic duct. Clamp and cut off the cystic duct near the gallbladder's neck with a Hemo-lock clamp. The cystic artery was found medial posterior side of the cystic duct. Clamp and cut off the cystic artery with Hemo-lock clamp. Pull the gallbladder's neck upward and remove the gallbladder by anterograde resection with an ultrasonic knife. The assistant assisted in dragging the gallbladder and the liver bed to keep a certain tension. The intact gallbladder was put into the specimen bag and removed. Bleeding and bile leakage was carefully checked, and the gallbladder bed was coagulated. The operating instruments were withdrawn from the patient's abdominal cavity after checking the instruments and the gauze. The pneumoperitoneum was exsufflated and the incisions were closed.

During the operation, the assembly time, intraoperative blood loss, operation time, operation success rate, and the adjacent organ and vascular injury caused by the failure of the tested system were recorded. Pain score was analyzed 24±2 hours after the surgery. The vital signs (temperature, pulse, respiration, blood pressure) were measured on the 3rd day postoperatively. Meanwhile, the routine blood test (red blood cells, white blood cells and neutrophils, platelet, hemoglobin), liver and renal function (ALT, AST, TP, ALB, GLU, TBIL, BUN, and CREA), the electrolyte (K, Na, Cl, Ca), blood sugar, and color ultrasound of liver, gallbladder, pancreas and spleen were checked. Operating surgeons filled in the satisfaction questionnaire postoperatively. Furthermore, the patients' postoperative condition changes, postoperative medication, the first postoperative anal exhaust, postoperative complications, and resident time were also recorded. All the patients were followed up by telephone at 30±5 days postoperatively to evaluate the incidncee of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* from 18 to 65 years old;
* patients with acute or chronic cholecystitis, gallstone, gallbladder polyp and other benign gallbladder diseases;
* BMI was 18-30 kg/m2;
* the American Society of Anesthesiologists (ASA) classification was I, II, or III.

Exclusion Criteria:

* women in pregnancy or lactation;
* A history of epilepsy or mental illness;
* Previous relevant operation history;
* Patients with a severe cardiovascular and cerebrovascular disease with New York Heart Association (NYHA) classification III-IV and pulmonary insufficiency who cannot tolerate the operation;
* Liver cirrhosis, kidney failure and other severe liver and kidney dysfunction (ALT and AST exceeded 3 times of the upper limit of normal value, Cr exceeded 1.5 times of the upper limit of normal value).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Success rate of the surgery | after the study is completed, up to 14 months
  the proportion of patients with successful operation in all participating patients in the experimental or control group

SECONDARY OUTCOMES:
assembly time | after the robot is assembled, all data will be collected within 14 months
  The assembly time extends from the time the robot starts to the time the trocar is connected to the robot arm.
operation time | after the procedure is completed, all data will be collected within 14 months
  The operation time extends from the time the robot assembles are finished, and the operation begins till the incision is sutured.
blood loss | after the procedure is completed, all data will be collected within 14 months
  Intraoperative blood loss is the total amount of blood loss from the beginning of the operation (after the robot was assembled) to the incision is sutured.
Time to first flatus | after the intestinal function revival of the patients, all data will be collected within 14 months
  Time to first flatus is the patients' first anal exhaust after the operation.
The hospital stay | from the admission to the discharge, all data will be collected within 14 months
  The hospital stay is the total number of days from the admission to the discharge of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Guo, MD, Study Chair — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Case record form of the patients will be shared within six months after the trial complete
Supporting Information: CSR
Time Frame: Case record form of the patients will be shared within six months after the trial complete

REFERENCES:
- [Background] Asad U, Wang CF, Jones MW. Laparoscopic Cholecystectomy. 2025 Jul 2. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448145/ PMID 28846328
- [Background] Abdel Raheem A, Troya IS, Kim DK, Kim SH, Won PD, Joon PS, Hyun GS, Rha KH. Robot-assisted Fallopian tube transection and anastomosis using the new REVO-I robotic surgical system: feasibility in a chronic porcine model. BJU Int. 2016 Oct;118(4):604-9. doi: 10.1111/bju.13517. Epub 2016 May 26. PMID 27123543
- [Background] Alli VV, Yang J, Xu J, Bates AT, Pryor AD, Talamini MA, Telem DA. Nineteen-year trends in incidence and indications for laparoscopic cholecystectomy: the NY State experience. Surg Endosc. 2017 Apr;31(4):1651-1658. doi: 10.1007/s00464-016-5154-9. Epub 2016 Sep 7. PMID 27604366
- [Background] Breitenstein S, Nocito A, Puhan M, Held U, Weber M, Clavien PA. Robotic-assisted versus laparoscopic cholecystectomy: outcome and cost analyses of a case-matched control study. Ann Surg. 2008 Jun;247(6):987-93. doi: 10.1097/SLA.0b013e318172501f. PMID 18520226
- [Background] Csikesz NG, Singla A, Murphy MM, Tseng JF, Shah SA. Surgeon volume metrics in laparoscopic cholecystectomy. Dig Dis Sci. 2010 Aug;55(8):2398-405. doi: 10.1007/s10620-009-1035-6. Epub 2009 Nov 13. PMID 19911275
- [Background] Fanfani F, Monterossi G, Fagotti A, Rossitto C, Gueli Alletti S, Costantini B, Gallotta V, Selvaggi L, Restaino S, Scambia G. The new robotic TELELAP ALF-X in gynecological surgery: single-center experience. Surg Endosc. 2016 Jan;30(1):215-21. doi: 10.1007/s00464-015-4187-9. Epub 2015 Apr 4. PMID 25840895
- [Background] Heemskerk J, van Dam R, van Gemert WG, Beets GL, Greve JW, Jacobs MJ, Bouvy ND. First results after introduction of the four-armed da Vinci Surgical System in fully robotic laparoscopic cholecystectomy. Dig Surg. 2005;22(6):426-31. doi: 10.1159/000091445. Epub 2006 Feb 10. PMID 16479111
- [Background] Huang Y, Chua TC, Maddern GJ, Samra JS. Robotic cholecystectomy versus conventional laparoscopic cholecystectomy: A meta-analysis. Surgery. 2017 Mar;161(3):628-636. doi: 10.1016/j.surg.2016.08.061. Epub 2016 Dec 20. PMID 28011011
- [Background] Li J, Zhu S, Juan J, Yi B. Preliminary exploration of robotic complete mesocolic excision for colon cancer with the domestically produced Chinese minimally invasive Micro Hand S surgical robot system. Int J Med Robot. 2020 Dec;16(6):1-8. doi: 10.1002/rcs.2148. Epub 2020 Sep 11. PMID 32865308
- [Background] Luo D, Liu Y, Zhu H, Li X, Gao W, Li X, Zhu S, Yu X. The MicroHand S robotic-assisted versus Da Vinci robotic-assisted radical resection for patients with sigmoid colon cancer: a single-center retrospective study. Surg Endosc. 2020 Aug;34(8):3368-3374. doi: 10.1007/s00464-019-07107-z. Epub 2019 Sep 3. PMID 31482355
- [Background] Melling N, Barr J, Schmitz R, Polonski A, Miro J, Ghadban T, Wodack K, Izbicki J, Zani S, Perez D. Robotic cholecystectomy: first experience with the new Senhance robotic system. J Robot Surg. 2019 Jun;13(3):495-500. doi: 10.1007/s11701-018-0877-3. Epub 2018 Sep 27. PMID 30264180
- [Background] Morelli L, Di Franco G, Lorenzoni V, Guadagni S, Palmeri M, Furbetta N, Gianardi D, Bianchini M, Caprili G, Mosca F, Turchetti G, Cuschieri A. Structured cost analysis of robotic TME resection for rectal cancer: a comparison between the da Vinci Si and Xi in a single surgeon's experience. Surg Endosc. 2019 Jun;33(6):1858-1869. doi: 10.1007/s00464-018-6465-9. Epub 2018 Sep 24. PMID 30251144
- [Background] Rassweiler JJ, Autorino R, Klein J, Mottrie A, Goezen AS, Stolzenburg JU, Rha KH, Schurr M, Kaouk J, Patel V, Dasgupta P, Liatsikos E. Future of robotic surgery in urology. BJU Int. 2017 Dec;120(6):822-841. doi: 10.1111/bju.13851. Epub 2017 Apr 22. PMID 28319324
- [Background] Strosberg DS, Nguyen MC, Muscarella P 2nd, Narula VK. A retrospective comparison of robotic cholecystectomy versus laparoscopic cholecystectomy: operative outcomes and cost analysis. Surg Endosc. 2017 Mar;31(3):1436-1441. doi: 10.1007/s00464-016-5134-0. Epub 2016 Aug 5. PMID 27495346
- [Background] Su M, Wang J, Li Z, Luo Z, Yuan S, Chen G, Liao Z, He C. [A New Micro-traumatic Laparoscopic Surgery Robot System]. Zhongguo Yi Liao Qi Xie Za Zhi. 2019 May 30;43(3):165-169. doi: 10.3969/j.issn.1671-7104.2019.03.003. Chinese. PMID 31184070
- [Background] Tang CL, Schlich T. Surgical Innovation and the Multiple Meanings of Randomized Controlled Trials: The First RCT on Minimally Invasive Cholecystectomy (1980-2000). J Hist Med Allied Sci. 2017 Apr 1;72(2):117-141. doi: 10.1093/jhmas/jrw027. PMID 27667536
- [Background] Yao Y, Liu Y, Li Z, Yi B, Wang G, Zhu S. Chinese surgical robot micro hand S: A consecutive case series in general surgery. Int J Surg. 2020 Mar;75:55-59. doi: 10.1016/j.ijsu.2020.01.013. Epub 2020 Jan 23. PMID 31982634
- [Background] Yi B, Wang G, Li J, Jiang J, Son Z, Su H, Zhu S. The first clinical use of domestically produced Chinese minimally invasive surgical robot system "Micro Hand S". Surg Endosc. 2016 Jun;30(6):2649-55. doi: 10.1007/s00464-015-4506-1. Epub 2015 Aug 21. PMID 26293795
- [Background] Yi B, Wang G, Li J, Jiang J, Son Z, Su H, Zhu S, Wang S. Domestically produced Chinese minimally invasive surgical robot system "Micro Hand S" is applied to clinical surgery preliminarily in China. Surg Endosc. 2017 Jan;31(1):487-493. doi: 10.1007/s00464-016-4945-3. Epub 2016 May 18. PMID 27194259
- [Background] Zeng Y, Wang G, Liu Y, Li Z, Yi B, Zhu S. The "Micro Hand S" Robot-Assisted Versus Conventional Laparoscopic Right Colectomy: Short-Term Outcomes at a Single Center. J Laparoendosc Adv Surg Tech A. 2020 Apr;30(4):363-368. doi: 10.1089/lap.2019.0714. Epub 2020 Feb 3. PMID 32013727